CLINICAL TRIAL: NCT04134104
Title: Incidence of The Bowel, Bladder, and Sexual Dysfunction Following Surgery for Colorectal Malignancy
Status: Completed | Type: Observational
Sponsor: National Academy of Medical Sciences, Nepal (Other Government)
Responsible Party: Principal Investigator, Nabin Pokharel, Assistant Professor/ Senior Medical Officer, National Academy of Medical Sciences, Nepal
Other Study IDs: 1145
Record Dates: First submitted 2019-09-17; First posted 2019-10-21 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Bowel Dysfunction; Bladder Dysfunction; Sexual Dysfunction; Colorectal Surgery
MeSH Terms: conditions — Intestinal Diseases; Sexual Dysfunction, Physiological | interventions — Surgical Procedures, Operative; Low Density Lipoprotein Receptor-Related Protein-1

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Bowel, Bladder, and Sexual Dysfunction group: Out of 38 patients included for surgery 12 were excluded due to poor follow up and those patients who underwent upfront surgery. Only 26 patients were included in the study. There were 20 (76.9%) males and 6 (23.1%) females respectively. The mean age of the patient was 43.577yrs (26-75) and mean BMI was 20.78. The number of patients that underwent LAR was 24 (92.30%) and those who underwent APR were 2( 7.6%) after neoadjuvant chemoradiotherapy respectively.
  Interventions: Procedure: Surgery for Colorectal malignant diseases either LAR or APR

INTERVENTIONS:
Procedure: Surgery for Colorectal malignant diseases either LAR or APR — Patients following LAR or APR were observed for the Bowel, Bladder, and Sexual Dysfunction

SUMMARY:
Colorectal cancer is the second most common cancer by the site in Europe and the third most common cancer in the USA with high morbidity and mortality. Survival after the treatment has improved over the past few decades as a result of early diagnosis, radiotherapy, and advances in surgical techniques such as abdominoperineal resection (APR), low anterior resection (LAR) and total mesorectal excision (TME). These innovative surgeries are the current standard treatment for the mid and the low rectal cancers which avoids the permanent colostomy. It is very difficult to find out the incidence of the bowel, bladder and sexual dysfunction of patients either because they are embarrassed or because they do not relate their symptoms to rectal cancer treatment. This article reports the incidence of the bowel, bladder and sexual dysfunction following surgery for rectal cancer from the National Academy of Medical Sciences, Bir Hospital, a tertiary level hospital.

DETAILED DESCRIPTION:
It was a cross-sectional study at Bir Hospital and the duration of the study was from December 2014 to December 2017. Here, all the patients who underwent LAR and APR following neoadjuvant chemoradiotherapy were included. And, all the patients with recurrence after surgery, lost to follow up, benign disease, who did not undergo neoadjuvant chemoradiotherapy, and who underwent trans-anal excision were excluded from the study. In our study, the independent variable will be the type of surgery done for colorectal malignant disease. And the dependent variables will be the postoperative complications in the form of immediate and delayed complications. Immediate could be infectious or non-infectious complications and delayed (long term) complications could be bowel, bladder, and sexual dysfunction respectively.

Data collection was done using structured Performa that included all the demographic parameters, examination findings which included the data regarding neoadjuvant chemoradiotherapy and type of surgery (LAR and APR) were included. The laboratory parameters were also included. All the operative and post-operative details were included regarding bowel, bladder, and sexual dysfunction. And validated tools were used to calculate and analyze data.

LARS Score Questionnaire: The aim of this questionnaire was to assess the bowel function using a validated questionnaire.6 The LARS consists of five questions and can be used to generate an overall score that translates into no LARS (score 0-20), minor LARS (21-29), and major LARS (30-42) respectively.

IPSS Questionnaire: Assessment of bladder dysfunction was assessed by the validated questionnaire of International Prostatic Symptoms Score (IPSS) for bladder dysfunction.8 For the evaluation of preoperative and postoperative bladder function, a urologic history and residual urine volume measurements by ultrasound were done.

Sexual Function Evaluation: In the early period after surgery sexual function was measured using the validated questionnaire - the International Index of Female Sexual Function (IFSF) for females and the International Index of Erectile Function (IIEF) for males. These tools helped to assess the impact of a specific treatment modality by evaluating different sexual function domains. Our study group was small, so we did not classify the groups into mild, moderate, and severe dysfunction groups. We did the overall long term assessment of the patients who came for the follow-up. These specific questionnaires were asked and the assessment was done for the overall dysfunctions.

Ethics: The study was approved by the institutional ethical committee- "IRB of NAMS, Bir Hospital" and written consent was obtained from all of the patients.

Statistics: All the data were entered in SPSS version 16 and then statistical analysis was done. Type of surgery, the status of neoadjuvant chemoradiotherapy, and the postoperative outcomes were studied respectively. Correlation and logistic regression statistic tools were used. A comprehensive literature search published in English was done until 2019 using Hinari, PubMed, and Cochrane Library.

ELIGIBILITY:
Inclusion Criteria:

1) All the patients who underwent LAR and APR following neoadjuvant chemoradiotherapy.

Exclusion Criteria:

1. All the patients with recurrence after surgery,
2. Lost to follow up,
3. Benign disease,
4. Patients who did not undergo neoadjuvant chemoradiotherapy, and
5. Patients who underwent trans-anal excision.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: It was a cross-sectional study at Bir Hospital and the duration of the study was from December 2014 to December 2017. Out of 38 patients included for surgery 12 were excluded due to poor follow up and those patients who underwent upfront surgery. Only 26 patients were included in the study. There were 20 (76.9%) males and 6 (23.1%) females respectively. The mean age of the patient was 43.577yrs (26-75) and mean BMI was 20.78. The number of patients that underwent LAR was 24 (92.30%) and those who underwent APR were 2( 7.6%) after neoadjuvant chemoradiotherapy respectively. Immediate could be infectious or non-infectious complications and delayed (long term) complication could be bowel, bladder, and sexual dysfunction respectively.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Bowel Dysfunction | 6 months
  Self reported urgency, fecal incontinence (either flatus or stool), difficulty in the evacuation. It is calculated using LARS Score Questionnaire which consists of five questions and can be used to generate an overall score that translates into no LARS (score 0-20), minor LARS (21-29), and major LARS (30-42) respectively.
Bladder Dysfunction | 6 months
  Self reported Weak urinary stream, stress incontinence, difficulty in postponing urination, dysuria. Assessment of bladder dysfunction was done by the validated questionnaire of International Prostatic Symptoms Score (IPSS) for bladder dysfunction.
Sexual Dysfunction | 6 months
  Self reported no sexual desire, unable to attain erection, unable to ejaculate, dyspareunia. The International Index of Female Sexual Function (IFSF) for females and the International Index of Erectile Function (IIEF) for males.

CONTACTS AND LOCATIONS:
Overall Officials: Nabin Pokharel, MCh, Principal Investigator — Bir Hospital; Gaurav Katwal, MS, Principal Investigator — Bir Hospital; Subodh K Adhikari, MS, Study Director — Bir Hospital

IPD SHARING:
Plan to Share IPD: Yes
If other researchers are interested in the IPD of our research. They can ask us through our email. We will provide the IPD.
Supporting Information: Study Protocol, SAP
Time Frame: It can be provided any time if asked via email.
Access Criteria: The interested researcher should contact the corresponding author.

REFERENCES:
- [Background] Juul T, Ahlberg M, Biondo S, Espin E, Jimenez LM, Matzel KE, Palmer GJ, Sauermann A, Trenti L, Zhang W, Laurberg S, Christensen P. Low anterior resection syndrome and quality of life: an international multicenter study. Dis Colon Rectum. 2014 May;57(5):585-91. doi: 10.1097/DCR.0000000000000116. PMID 24819098
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2019. CA Cancer J Clin. 2019 Jan;69(1):7-34. doi: 10.3322/caac.21551. Epub 2019 Jan 8. PMID 30620402
- [Background] Hawkins AT, Albutt K, Wise PE, Alavi K, Sudan R, Kaiser AM, Bordeianou L; Continuing Education Committee of the SSAT. Abdominoperineal Resection for Rectal Cancer in the Twenty-First Century: Indications, Techniques, and Outcomes. J Gastrointest Surg. 2018 Aug;22(8):1477-1487. doi: 10.1007/s11605-018-3750-9. Epub 2018 Apr 16. PMID 29663303
- [Background] Yeom SS, Park IJ, Jung SW, Oh SH, Lee JL, Yoon YS, Kim CW, Lim SB, Kim N, Yu CS, Kim JC. Outcomes of patients with abdominoperineal resection (APR) and low anterior resection (LAR) who had very low rectal cancer. Medicine (Baltimore). 2017 Oct;96(43):e8249. doi: 10.1097/MD.0000000000008249. PMID 29068989
- [Background] Heald RJ, Ryall RD. Recurrence and survival after total mesorectal excision for rectal cancer. Lancet. 1986 Jun 28;1(8496):1479-82. doi: 10.1016/s0140-6736(86)91510-2. PMID 2425199
- [Background] Juul T, Ahlberg M, Biondo S, Emmertsen KJ, Espin E, Jimenez LM, Matzel KE, Palmer G, Sauermann A, Trenti L, Zhang W, Laurberg S, Christensen P. International validation of the low anterior resection syndrome score. Ann Surg. 2014 Apr;259(4):728-34. doi: 10.1097/SLA.0b013e31828fac0b. PMID 23598379
- [Background] Adam JP, Denost Q, Capdepont M, van Geluwe B, Rullier E. Prospective and Longitudinal Study of Urogenital Dysfunction After Proctectomy for Rectal Cancer. Dis Colon Rectum. 2016 Sep;59(9):822-30. doi: 10.1097/DCR.0000000000000652. PMID 27505110
- [Background] Rosen R, Brown C, Heiman J, Leiblum S, Meston C, Shabsigh R, Ferguson D, D'Agostino R Jr. The Female Sexual Function Index (FSFI): a multidimensional self-report instrument for the assessment of female sexual function. J Sex Marital Ther. 2000 Apr-Jun;26(2):191-208. doi: 10.1080/009262300278597. PMID 10782451
- [Background] Rosen RC, Riley A, Wagner G, Osterloh IH, Kirkpatrick J, Mishra A. The international index of erectile function (IIEF): a multidimensional scale for assessment of erectile dysfunction. Urology. 1997 Jun;49(6):822-30. doi: 10.1016/s0090-4295(97)00238-0. PMID 9187685
- [Background] Bregendahl S, Emmertsen KJ, Lous J, Laurberg S. Bowel dysfunction after low anterior resection with and without neoadjuvant therapy for rectal cancer: a population-based cross-sectional study. Colorectal Dis. 2013 Sep;15(9):1130-9. doi: 10.1111/codi.12244. PMID 23581977
- [Background] Keane C, Wells C, O'Grady G, Bissett IP. Defining low anterior resection syndrome: a systematic review of the literature. Colorectal Dis. 2017 Aug;19(8):713-722. doi: 10.1111/codi.13767. PMID 28612460
- [Background] Kupsch J, Jackisch T, Matzel KE, Zimmer J, Schreiber A, Sims A, Witzigmann H, Stelzner S. Outcome of bowel function following anterior resection for rectal cancer-an analysis using the low anterior resection syndrome (LARS) score. Int J Colorectal Dis. 2018 Jun;33(6):787-798. doi: 10.1007/s00384-018-3006-x. Epub 2018 Mar 15. PMID 29541896
- [Background] Lange MM, Maas CP, Marijnen CA, Wiggers T, Rutten HJ, Kranenbarg EK, van de Velde CJ; Cooperative Clinical Investigators of the Dutch Total Mesorectal Excision Trial. Urinary dysfunction after rectal cancer treatment is mainly caused by surgery. Br J Surg. 2008 Aug;95(8):1020-8. doi: 10.1002/bjs.6126. PMID 18563786
- [Background] Doeksen A, Gooszen JA, van Duijvendijk P, Tanis PJ, Bakx R, Slors JF, van Lanschot JJ. Sexual and urinary functioning after rectal surgery: a prospective comparative study with a median follow-up of 8.5 years. Int J Colorectal Dis. 2011 Dec;26(12):1549-57. doi: 10.1007/s00384-011-1288-3. Epub 2011 Sep 16. PMID 21922200
- [Background] Junginger T, Kneist W, Heintz A. Influence of identification and preservation of pelvic autonomic nerves in rectal cancer surgery on bladder dysfunction after total mesorectal excision. Dis Colon Rectum. 2003 May;46(5):621-8. doi: 10.1007/s10350-004-6621-2. PMID 12792438
- [Background] Hendren SK, O'Connor BI, Liu M, Asano T, Cohen Z, Swallow CJ, Macrae HM, Gryfe R, McLeod RS. Prevalence of male and female sexual dysfunction is high following surgery for rectal cancer. Ann Surg. 2005 Aug;242(2):212-23. doi: 10.1097/01.sla.0000171299.43954.ce. PMID 16041212
- [Background] Bruheim K, Guren MG, Dahl AA, Skovlund E, Balteskard L, Carlsen E, Fossa SD, Tveit KM. Sexual function in males after radiotherapy for rectal cancer. Int J Radiat Oncol Biol Phys. 2010 Mar 15;76(4):1012-7. doi: 10.1016/j.ijrobp.2009.03.075. Epub 2009 Oct 31. PMID 19880263
- [Background] Vironen JH, Kairaluoma M, Aalto AM, Kellokumpu IH. Impact of functional results on quality of life after rectal cancer surgery. Dis Colon Rectum. 2006 May;49(5):568-78. doi: 10.1007/s10350-006-0513-6. PMID 16583289
- See also: Cancer incidence and mortality patterns in Europe: Estimates for 40 countries and 25 major cancers in 2018 — https://doi.org/10.1016/j.ejca.2018.07.005
- See also: A prospective study of sexual and urinary function before and after total mesorectal excision — http://dx.doi.org/10.1007/s00384-016-2549-y